CLINICAL TRIAL: NCT02985190
Title: A Phase II Study of Efficacy and Tolerance of Azacitidine (AZA) In MDS-associated Steroid Dependent/Refractory Systemic Auto-immune and Inflammatory Disorders (SAID)
Brief Title: A Study of Azacitidine in Myelodysplastic Syndrome (MDS) Associated to Systemic Auto-immune and Inflammatory Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Groupe Francophone des Myelodysplasies (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GFM-AZA-SAID; 2016-000918-30 (EudraCT Number)
Record Dates: First submitted 2016-11-07; First posted 2016-12-07 (Estimated); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: MDS; Systemic Autoimmune Diseases
Keywords: Azacitidine; MDS; Systemic auto-immune and inflammatory disorders
MeSH Terms: interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Azacitidine 75mg/m²/day (Experimental): Azacitidine 75mg/m²/j subcutaneously daily for 7 days every 4 weeks for a minimum of 6 cycles (unless overt disease progression, especially to Acute Myeloid Leukemia (AML) occure before 6 cycles) Azacitidine will be continued after 6 cycles
  * in patients with hematological response of myelodysplastic syndrome to azacitidine according to IWG2006 criteria by 6 cycles (Complete Response (CR), Partial Response (PR), marrow Complete Response (CRm), stable disease with Hematological Improvment (HI)), for another 6 cycles
  * in patients with complete or partial response of Systemic Auto-Immune Disorders (SAID) after 6 cycles of Azacitidine, even if Myelodysplastic Syndrome remains only stable per IWG2006 criteria
  Interventions: Drug: Azacitidine

INTERVENTIONS:
Drug: Azacitidine — Azacitidine at 75mg/m²/j for 7 days.
  Other Names: Vidaza

SUMMARY:
This study is a phase II of effcicacy and tolerance of azacitidine in patients with myelodysplatic syndrome and steroid dependent or resistent systemic auto-immune and inflammatory disorders

DETAILED DESCRIPTION:
This trial will be a prospective French nationwide study analyzing the effect of treatment with azacitidine in patients with MDS-associated SAID with steroid dependence and/or resistance, and its correlation with possible changes in immunological parameters

ELIGIBILITY:
Inclusion Criteria:

* Must understand and voluntarily sign the informed consent form
* Age 18 years at the time of signing the informed consent form
* Must be able to adhere to the study visit schedule and other protocol requirements
* MDS or CMML or AML with 20-30% marrow blasts using 2008 WHO classification, with any of the following characteristics :

  1. IPSS intermediate 2 or high, including AML with 20 to 30% marrow blasts and CMML with WBC<13G/L and marrow blasts >10%,
  2. IPSS low or int 1 in need of treatment (transfusion dependent anemia resistant to ESAs and/or platelets below 30 G/l or below 50 G/l with bleeding or platelet transfusion requirement, and/or ANC < 0.5 G/l with infectious complications)
  3. Documented (by cytogenetic or molecular analysis) MDS /CMML not meeting those criteria, but with at least one significant cytopenia (Hb <10 g/dl, platelets <50G/l, ANC <1 G/l). In this situation, the underlying SAID should be severe and have resisted to a second line treatment (following steroids), if such treatment can be proposed for this particular SAID. Those cases should be discussed prior to inclusion with the trial sponsors complications)
* SAID-associated with MDS defined according to usual international criteria for each SAID (ie ACR criteria for systemic lupus, Chapel Hill classification for systemic vasculitis, etc…)
* Steroid dependence and/or resistance of SAID (steroid dependence being defined as the impossibility to decrease steroids during at least 2 months below 15 mg/day; steroid resistance as no response of SAID to at least 1 mg/kg/day of prednisone equivalent during one month)
* Ineligibility for allogeneic stem cell transplantation during the following 12 months
* Wash-out at least 6 months since a previous treatement with Lenalidomide
* No previous use of hypomethylating agents
* Life expectancy ≥ 6 months
* Adequate liver function (serum transaminases ≤ 3N)
* Adequate renal function (creatinine clearance with MDRD formula > 30 ml/min)
* Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must :

  * Have a negative serum or urine pregnancy test within 2 weeks prior to beginning treatment on this study. Lactating patients are excluded.
  * Agree to use, and to be able to comply with, effective contraception without interruption, 4 weeks before starting study drug throughout the entire duration study drug therapy (including doses interruptions) and for 3 months after the end of the study drug therapy.
* Male patients must :

  * Agree the need for the use of a condom if engaged in sexual activity with a woman of childbearing potential during the entire period of treatment, even if disruption of treatment and during 3 months after end of treatment.
  * Agree to learn about the procedures for preservation of sperm before starting treatment.

Exclusion Criteria:

* IPSS low and intermediate-1 not meeting the criteria described above
* Creatinine clearance with MDRD formula < 30 ml/min
* Serum total bilirubin, or serum transaminases > 3.0 x upper limit of normal (ULN) (except for unconjugated hyperbilirubinemia due to Gilbert's disease or secondary to MDS)
* Known hypersensitivity to the active substance or to any of the excipients of AZA
* History of severe congestive heart failure, clinically unstable cardiac or pulmonary disease
* Previous treatment with hypomethylating agents
* Life-expectancy of less than six months because of another debilitating disease
* Uncontrolled invasive fungal infection at time of registration or active serious infection not controlled by oral or intravenous antibiotics
* Known positive for HIV or acute infectious hepatitis, type B or C
* Any serious medical condition or psychiatric illness that will prevent the subject from signing the informed consent form or will place the subject at unacceptable risk if he/she participates in the study.
* Active cancer or prior history of malignancy other than MDS (except basal cell or squamous cell carcinoma or carcinoma in situ of the cervix or breast) unless the subject has been free of disease for ≥ 3 years
* Pregnant or lactating females
* No affiliation to an insurance system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-01-26 (Actual); Primary Completion 2021-09-02 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Overall response rate of Myelodysplastic syndrome and systemic autoimmune and inflammatory diseases (SAID) | 6 months
  Overall response rate (including partial and complete response) of systemic autoimmune and inflammatory diseases associated with Myelodysplastic syndrome after 6 cycles of azacitidine

SECONDARY OUTCOMES:
Number of participants with treament-related adverse events as assessed by CTCAE v4.0 | up to 52 weeks
  Number of participants with treament-related adverse events as assessed by CTCAE v4.0

OTHER OUTCOMES:
Overall survival | 24 months
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Arsene MEKINIAN, MD, Principal Investigator — Saint Antoine Hospital; Olivier FAIN, PHD, Principal Investigator — Saint Antoine Hospital; Pierre FENAUX, PHD, Study Director — Saint-Louis Hospital, Paris, France
Locations (59):
- France (59):
  - CHU Amiens, Amiens
  - CHU d'Angers, Angers
  - Centre hospitalier Victor Dupouy, Argenteuil
  - CH Henri Duffaut d'Avignon, Avignon
  - Centre hospitalier de la Côte Basque, Bayonne
  - Hôpital Nord Franche-Comté, Belfort
  - Hôpital Avicenne, Bobigny
  - Centre Hospitalier de Boulogne Sur Mer, Boulogne-sur-Mer
  - CHRU de Brest - Hôpital Morvan, Brest
  - CHU Côte de Nacre, Caen
  - CH René Dubos, Cergy-Pontoise
  - Centre Hospitalier William Morey, Chalon-sur-Saône
  - CHU Estaing, Clermont-Ferrand
  - CHSF Gilles de Corbeil, Corbeil-Essonnes
  - CHU Henri Mondor, Créteil
  - CHU François Mitterrand, Dijon
  - CHU de Grenoble, Grenoble
  - Groupe Hospitalier de la Rochelle Ré Aunis, La Rochelle
  - Clinique Victor Hugo - Centre Jean Bernard, Le Mans
  - CH Le Mans, Le Mans
  - Centre Hospitalier de Lens, Lens
  - Hôpital Saint Vincent de Paul, Lille
  - Hôpital Claude Huriez, Lille
  - CHRU de Limoges - Hôpital Dupuytren, Limoges
  - Institut Paoli Calmettes, Marseille
  - Centre Hospitalier de Meaux, Meaux
  - CH de Mont de Marsan, Mont-de-Marsan
  - Clinique Beausoleil, Montpellier
  - CHRU de Montpellier - Service de Médecine Interne, Montpellier
  - CHU de Montpellier - Service d'hématologie Oncologie, Montpellier
  - CHU Nantes - Hôtel Dieu, Nantes
  - Centre Catherine de Sienne, Nantes
  - Centre Antoine Lacassagne, Nice
  - Hôpital Archet 1, Nice
  - CHU de Nîmes, Nîmes
  - CHR d'Orléans, Orléans
  - Hôpital Saint-Louis, Paris
  - Hôpital Saint Antoine - Service de Médecine Interne, Paris
  - Hôpital de La Pitié-Salpêtrière, Paris
  - Hôpital Saint Antoine - Service d'Hématologie Clinique, Paris
  - Hôpital Cochin, Paris
  - Hôpital Necker, Paris
  - Centre Hospitalier Joffre, Perpignan
  - CHU de Haut-Lévèque, Pessac
  - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - CHU de Poitiers, Poitiers
  - Centre Hospitalier Annecy Genevois, Pringy
  - CHU de Reims, Reims
  - Hôpital PONTCHAILLOU, Rennes
  - Centre Hospitalier de Rochefort, Rochefort
  - Centrer Hospitalier de Roubaix, Roubaix
  - Centre Henri Becquerel, Rouen
  - CH Yves Le Foll, Saint-Brieuc
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - IUCT Oncopole, Toulouse
  - Hôpital Bretonneau, Tours
  - Centre Hospitalier de Troyes, Troyes
  - CH Valence, Valence
  - CHU Brabois, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Boy M, Bisio V, Zhao LP, Guidez F, Schell B, Lereclus E, Henry G, Villemonteix J, Rodrigues-Lima F, Gagne K, Retiere C, Larcher L, Kim R, Clappier E, Sebert M, Mekinian A, Fain O, Caignard A, Espeli M, Balabanian K, Toubert A, Fenaux P, Ades L, Dulphy N. Myelodysplastic Syndrome associated TET2 mutations affect NK cell function and genome methylation. Nat Commun. 2023 Feb 3;14(1):588. doi: 10.1038/s41467-023-36193-w. PMID 36737440